CLINICAL TRIAL: NCT01800487
Title: The Efficacy of Silymarin on the Prevention of Hepatotoxicity From Antituberculosis Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Abhasnee Sobhonslidsuk, Associate professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ramathibodi_silymarin
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Tuberculosis
Keywords: Drug-induced liver injury; Tuberculosis; Silymarin
MeSH Terms: conditions — Tuberculosis; Chemical and Drug Induced Liver Injury | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- silymarin (Active Comparator): Silymarin 140 mg three times a day for 4 weeks
  Interventions: Drug: silymarin
- placebo (Placebo Comparator): Placeo
  1 tab three times a day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: silymarin — 140 mg three times a day for 4 weeks
  Arms: silymarin
Drug: Placebo — Placebo (silymarin) 1 tab three times a day for 4 weeks
  Arms: placebo

SUMMARY:
Hepatitis is one of the most common adverse effect from anti-tuberculosis. Silymarin showed its efficacy to decreased serum alanine transaminase enzyme in animal models from recent study. No confirmed this efficacy was performed in human.

A prospective, double-blind, placebo-controlled trial was carried out according to Good Clinical Practice Guideline. This study is to define the efficacy of silymarin to prevent hepatotoxicity from anti-tuberculosis drugs. Informed consent is obtained prior to the study. New patients diagnosed with tuberculosis are enrolled. Patients with liver diseases, current alcohol drinking more than 20 g/day, regular use of herbal or other potential hepatotoxic drugs are excluded. Patients are treated with a standard regimen of four anti-tuberculosis therapy. They will randomize to receive either placebo or silymarin (140 mg) thrice daily. Liver function test (LFT) and clinical changes are assessed at 2- and 4-week after initiation of the treatment. DILI from anti-tuberculosis drugs ('atb-DILI') is defined as: i) a rise of alanine aminotransferase (ALT) to 2 times above normal upper limit, or ii) an elevation of total bilirubin more than 2 mg/dl with or without ALT elevation. The study endpoints are the level of ALT by week 4 and the number of patients who developed atb-DILI.

Statistical analysis is used to compare the differences in ALT and number of atb-DILI

DETAILED DESCRIPTION:
- Prevention of antituberculosis-related drug induced liver injury with silymarin is investigated.

ELIGIBILITY:
Inclusion Criteria:

* tuberculosis cases
* treated with isoniazid, rifampicin, ethambutol and pyrazinamide

Exclusion Criteria:

* no known liver disease (HBV, HCV), and HIV infection
* normal ALT level before enrollment
* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The number of patients who develop drug-induced liver injury (DILI) at 4 weeks | 4 weeks
  DILI from anti-tuberculosis drugs ('atb-DILI') is defined as: i) a rise of alanine aminotransferase (ALT) to 2 times above normal upper limit, or ii) an elevation of total bilirubin more than 2 mg/dl with or without ALT elevation.

CONTACTS AND LOCATIONS:
Overall Officials: Abhasnee Sobhonslidsuk, MD, Study Director — Ramathibodi Hospital; Chote Luangchosiri, MD, Principal Investigator — Ramathibodi
Locations (1):
- Gastroenterology and Hepatology, Ramathibodi hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Luangchosiri C, Thakkinstian A, Chitphuk S, Stitchantrakul W, Petraksa S, Sobhonslidsuk A. A double-blinded randomized controlled trial of silymarin for the prevention of antituberculosis drug-induced liver injury. BMC Complement Altern Med. 2015 Sep 23;15:334. doi: 10.1186/s12906-015-0861-7. PMID 26400476